CLINICAL TRIAL: NCT01602276
Title: The Effect of Transcranial Direct Current Stimulation on Subcortical Brain Functioning
Brief Title: The Effect of tDCS on Subcortical Brain Functioning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty identifying appropriate patients
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00047863
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Brain Damage, Chronic
Keywords: Parkinson's disease; Lewy body dementia; Korsakoff's syndrome; Subcortical Dementia; Huntington's Disease
MeSH Terms: conditions — Brain Damage, Chronic; Parkinson Disease; Lewy Body Disease; Korsakoff Syndrome; Huntington Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Stimulation (Experimental): Transcranial direct current stimulation using Anodal or Cathodal stimulation over the area of interest
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)
- Sham Stimulation (Sham Comparator): Transcranial direct current stimulation (tDCS) that is ramped up and ramped down providing the sensation of tDCS without delivering the full amount of tDCS.
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation (tDCS) — Anodal, Cathodal or Sham tDCS

SUMMARY:
This research is being done to determine whether transcranial direct current stimulation (tDCS) can improve certain abilities related to cognition, emotion and/or physical functioning in individuals with subcortical brain damage.

DETAILED DESCRIPTION:
While cortical brain structures are thought to be responsible for higher level cognitive functioning (i.e., perception, thoughts, language, memory, attention, and processing), subcortical brain regions (i.e., amygdala, midbrain, hippocampus, and thalamus) are generally believed to be responsible for more fundamental bases of such functions. A significant fraction of the population suffer from disabling disorders and diseases (i.e., Parkinson's disease, subcortical dementia, hypoxic brain damage) that affect subcortical areas. Despite their prevalence, very little success has been achieved in treating such impairments effectively.

This study has two main goals. One is to examine the effect of stimulation on a variety of subcortical functions (i.e., level of alertness, mood, cognition, and motor responding). A second goal is to examine the effects of varying some of the stimulus parameters of tDCS, notably the placement of the electrodes and the duration and frequency of application of current.

Adult participants with a confirmed diagnosis of subcortical brain damage, as well as healthy adults will be randomly assigned to anodal and cathodal stimulation in a counterbalanced order, and both will engage in simple behavioral tasks and/or physiological monitoring. These tasks will be specific to the deficit of interest.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in the English language
* History of subcortical brain damage (patient group only)
* No known neurological or cognitive impairment (control group only)

Exclusion Criteria:

* Appreciable deficits in hearing
* Schizophrenia, bipolar disorder, or major depression (normal controls only)
* Any neurological disorder associated with cognitive impairment or neuroanatomic abnormality (normal controls only)
* Language-based learning disorder (normal controls only)
* Dementia or Mini-Mental State Exam <24 for normal control participants
* Any implanted metal device (precludes use of tDCS)
* Any implanted cardiac pacemaker

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Improvement in motor functioning | 1 month
Improvement in level of consciousness and alertness | 1 month
Improvement in cognitive functioning | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Barry Gordon, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Department of Neurology; Cognitive Neurology/Neuropsychology, Baltimore, Maryland, United States